CLINICAL TRIAL: NCT06985485
Title: Sequential Blinatumomab and Inotuzumab Ozogamicin Immunotherapy in Newly Diagnosed B-ALL Patients Unfit/Fit-Declined for Intensive Chemotherapy: A Prospective, Open-Label, Single-Arm Phase II Trial
Brief Title: Full-Course Immunotherapy Consolidation for Unfit or Fit B-ALL Who Decline Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Prof., The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZBALL03
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia; Immunotherapy; Blinatumomab; Inotuzumab Ozogamicin
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unfit and Fit-Decline B-ALL (Experimental): Unfit B-ALL patients are defined as whose physical conditions are unable to tolerate standard intensive chemotherapy regimens by investigators. Fit-decline B-ALL patients are defined as who have adequate physiological capacity but declined to undergo intensive chemotherapy. A low-intensity chemotherapy regimen combined with a sequential treatment regimen of blinatumomab and inotuzumab ozogamicin is implemented.
  Interventions: Drug: Blinatumomab and Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Blinatumomab and Inotuzumab Ozogamicin — Subjects who meet the study criteria during screening will receive induction therapy consisting of low-intensity chemotherapy combined with BiTE with or without TKIs. Regimen includes dexamethasone, vindesine, followed by blinatumomab dosed by body weight: pts ≥45 kg receive fixed dosing (9 µg/day days 1-7, 28 µg/day days 8-28), pts <45 kg receive BSA-adjusted dosing (5 µg/m²/day days 1-7, 15 µg/m²/day days 8-28). Philadelphia chromosome-positive ALL pts receive second-generation TKIs, with subsequent switch to third-generation TKIs upon resistance. If morphologic remission is not achieved after initial therapy, a salvage cycle with InO will be administered. Post-remission consolidation chemotherapy includes high-dose methotrexate followed by sequential immunotherapy: BiTE (per weight-stratified dosing), then after a 2-week break, InO (0.8 mg/m² on day 1), followed by another 2-week break.This sequence is repeated for 4 cycles.
  Other Names: Full-Course Immunotherapy

SUMMARY:
This trial is a non-blinded, single-center, open-label, single-arm clinical study to investigate a full-course immunotherapy regimen in Unfit or Fit B-cell acute lymphoblastic leukemia (B-ALL) patients who decline chemotherapy (Fit-Decline). The trial aims to explore the efficacy and safety of sequential blinatumomab and inotuzumab ozogamicin therapy. The primary endpoint is overall survival (OS), while secondary endpoints include complete remission rate(CRR)、Objective Response Rate(ORR)、Event-free survival(EFS)、Relapse-free survival(RFS)、Cumulative incidence of relapse(CIR)、Non-relapse mortality(NRM) and safety.

ELIGIBILITY:
Inclusion Criteria:

-

(1) Newly diagnosed B-cell acute lymphoblastic leukemia (B-ALL) patients aged ≥60 years, as per the NCCN 2024 guidelines.

(2) Newly diagnosed B-ALL patients aged ≥15 and <60 years who are unfit for intensive chemotherapy(Unfit), as per the NCCN 2024 guidelines, and have at least one of the following:

1. ECOG score ≥2.
2. Severe cardiac comorbidities (e.g., treated congestive heart failure, echocardiogram LVEF ≤50%, unstable angina).
3. Severe pulmonary comorbidities (e.g., DLCO ≤65%, FEV1 ≤65%).
4. Severe renal comorbidities (e.g., serum creatinine >2×upper limit of normal (ULN), creatinine clearance <45 mL/min by any formula).
5. Severe hepatic comorbidities (e.g., total bilirubin >1.5× ULN, AST/ALT/ALP >3.0× ULN).
6. Active infection unresponsive to antimicrobial therapy.
7. Cognitive impairment.
8. Other comorbidities contraindicating chemotherapy. (3) Newly diagnosed B-ALL patients aged ≥15 years who are physically fit and have normal organ function but refuse intensive chemotherapy for subjective reasons(Fit-Declined) (e.g., fear of toxicity, financial/social/psychological factors, preference for improving quality of life), as per the NCCN 2024 guidelines.

(4) Adequate major organ function:

1. Echocardiogram LVEF ≥40%.
2. creatinine clearance ≥30 mL/min by any formula.
3. ALT/AST ≤3× ULN, total bilirubin ≤2× ULN (excluding leukemia-related cases).
4. ≤Grade 1 dyspnea , oxygen saturation >91% without supplemental oxygen. (5) Ability to understand and voluntarily sign the informed consent form. (6) Life expectancy ≥3 months.

Exclusion Criteria:

1. Presence of extramedullary disease.
2. Concurrent other active or treatment-requiring malignancies.
3. Prior CD19/CD22-targeted therapy.
4. Use of immunosuppressive agents within 2 weeks before signing informed consent, or planned long-term immunosuppressive therapy after enrollment.
5. Active NYHA Class ≥3 heart disease.
6. Severe chronic liver disease (e.g., cirrhosis, nodular regenerative hyperplasia, active hepatitis [HBsAb-positive, HCVAb-positive]).

   * Occult or resolved HBV infection (defined as HBcAb-positive but HBsAg-negative) is allowed only if HBV DNA PCR is negative, with mandatory monthly HBV DNA monitoring and prophylactic antiviral therapy.
   * HCV antibody-positive patients are eligible only if HCV RNA PCR is negative.
   * History of severe or persistent VOD/SOS (veno-occlusive disease/sinusoidal obstruction syndrome).
7. Uncontrolled bacterial, fungal, viral, mycoplasma, or other infections as judged by the investigator, including HIV, syphilis, or SARS-CoV-2 infection.
8. Past/current CNS disorders (e.g., seizures, cerebrovascular events, dementia, cerebellar disease, CNS autoimmune diseases).
9. Primary immunodeficiency or active autoimmune disease.
10. History of severe immediate hypersensitivity to any study drugs.
11. Live vaccine receipt within 6 weeks before screening.
12. Psychiatric disorders or other conditions that may compromise compliance with study procedures, treatment, or monitoring.
13. Pregnant/breastfeeding women, or fertile patients not using contraception.
14. Any other condition deemed unsuitable for study participation by the investigator.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | 2 years
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.

SECONDARY OUTCOMES:
CR rate(CRR) | 2 years
  CR rate (CR defined as bone marrow blasts < 5% and no Auer rods, absence of extramedullary disease, ANC ≥ 1.0 × 109/L [1000/µL], platelet count ≥ 100 × 109/L [100,000/µL], and independence of RBC transfusions).
Objective Response Rate (ORR) | 2 years
  Objective response rate (ORR) is defined as the rate of CR, CRi (including complete remission with incomplete platelet recovery [CRp], PR, and MLFS.
Event-free survival(EFS) | 2 years
  Event-free survival (EFS) is defined as the time from the start of treatment until treatment failure, relapse from remission, or death from any cause, whichever occurs first.
Relapse-free survival(RFS) | 2 years
  Relapse-free survival(RFS) is the time from achievement of complete remission (CR) to the first documented relapse or death from any cause. Patients who die without evidence of relapse are typically censored at the last disease-free assessment.
Cumulative incidence of relapse(CIR) | 2 years
  It is measured the date from complete remission to hematological relapse or molecular relapse was recorded. Patients who had no relapse at the last follow-up were considered as censored data, and non-relapse death was regarded as a competing risk event.
Non-relapse mortality(NRM) | 2 years
  It is measured the probability of death attributable to treatment-related complications or comorbidities, excluding disease relapse/progression.

OTHER OUTCOMES:
immune function | 2 years
  To investigate the impact of the full-course sequential immunotherapy regimen on patients' immune function.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Li Xue, M.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China